CLINICAL TRIAL: NCT00421967
Title: Postoperative Analgesia After Total Knee Arthroplasty. A Comparison of Continuous Epidural Infusion and Wound Infiltration With Continuous Intraarticular Infusion
Brief Title: Postoperative Analgesia After Total Knee Arthroplasty
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Interim analysis
Sponsor: University of Aarhus (Other)
Responsible Party: Kjeld Soballe, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-004638-33.
Record Dates: First submitted 2007-01-12; First posted 2007-01-15 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-05

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Ketorolac; Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Ropivacaine, Ketorolac, adrenaline
- 2 (Active Comparator)
  Interventions: Drug: Ropivacaine Ketorolac

INTERVENTIONS:
Drug: Ropivacaine, Ketorolac, adrenaline — Infiltration: 150 ml Ropivacaine 2mg/ml added 1 ml Ketorolac 30 mg/ml and 0,5 ml Adrenaline 1 mg/ml Intraarticular infusion: 4 ml/h 384 mg Ropivacaine 60 mg Ketorolac
  Arms: 1
Drug: Ropivacaine Ketorolac — Epidural infusion: 4 ml/h 384 mg Ropivacaine I.V. Ketorolac 90 mg
  Arms: 2

SUMMARY:
Total knee arthroplasty (TKA) is associated with moderate to severe postoperative pain. Although epidural treatment provides good and reliable postoperative pain relief after THA, it may cause urinary retention, nausea, hypotension, diminished muscle control, and delayed mobilization.

The challenge of new analgesic regimes is to reduce the occurrence of side effects while maintaining adequate pain relief and maximum muscle control. A relatively new method to provide postoperative pain relief after TKA is local infiltration analgesia combined with single-shot injection(s) or continuous infusion of local anesthetics into the surgical site. As local infiltration analgesia combined with continuous intraarticular infusion compared with continuous epidural infusion has not been evaluated, our study was designed to determine whether this technique could enhance analgesia and improve patient outcome after TKA. This study compares continuous epidural infusion of Ropivacaine and intravenous Ketorolac with local infiltration analgesia with Ropivacaine, Ketorolac and Adrenaline combined with continuous intraarticular infusion of Ropivacaine and Ketorolac.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted consecutively to primary total knee arthroplasty.
* Provided informed consent

Exclusion Criteria:

* Fertile women with positive pregnancy test, nursing mothers, fertile women who do not use safe contraception
* Severe chronic neurogenic pain
* Medical treated diabetes
* Contraindications for spinal aesthesia and epidural analgesia
* Known hypersensitivity towards study drugs
* Rheumatoid arthritis
* Treatment with narcotics
* Treatment with antidepressants
* Severe obesity BMI>35
* Treatment with antacid
* Not able to speak and understand Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-01; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Analgésia consumption | 48 h

SECONDARY OUTCOMES:
Time to discharge
Cytokine level | 48 h
Pain scores VAS | 72 h
Side-effects | 72 h

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte V Christensen, M.D., Principal Investigator — Glostrup Hospital, Glostrup 2600, Denmark
Locations (1):
- Glostrup Hospital, Glostrup Municipality, Denmark